CLINICAL TRIAL: NCT01206790
Title: Immunological Changes Through Narrative Treatment of PTSD in Torture Victims
Brief Title: Immunological Changes Through Narrative Treatment of Post-Traumatic Stress Disorder (PTSD) in Torture Victims
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Iris-Tatjana Kolassa, Prof. Dr. Iris-Tatjana Kolassa, University of Ulm
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NET-2010-KN
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: PTSD
Keywords: PTSD; Narrative Exposure Therapy; torture victims; immune system
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Narrative Exposure Therapy (NET) (Experimental)
  Interventions: Behavioral: NET
- Waitinglist Control Group (No Intervention)

INTERVENTIONS:
Behavioral: NET — Narrative Exposure Therapy for traumatized survivors of organized violence
  Arms: Narrative Exposure Therapy (NET)

SUMMARY:
Posttraumatic stress disorder (PTSD) is associated with poor health, high health care utilization, and an increased risk for a variety of somatic, inflammatory and autoimmune diseases. Research, including our own findings, indicates immunological alterations in PTSD patients. The aim of this study is to investigate whether alterations in the immune system of PTSD patients are reversible through a trauma-specific short-term therapy (Narrative Exposure Therapy).

ELIGIBILITY:
Inclusion Criteria:

* PTSD diagnosis
* experiences of organized violence/torture

Exclusion Criteria:

* psychotic disorder
* chronic inflammatory diseases

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2009-06; Primary Completion 2011-05 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
PTSD diagnosis and severity score according to the Clinicians Administered PTSD Scale (CAPS) | 4 month after completion of treatment

SECONDARY OUTCOMES:
changes in immunological parameters | 4 months after completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Iris-Tatjana Kolassa, Prof. Dr., Principal Investigator — University of Ulm
Locations (1):
- University of Konstanz, Department of Psychology, Konstanz, Germany